CLINICAL TRIAL: NCT02106091
Title: A Pharmacodynamically-guided, Dose-escalation, Phase I Study to Assess the Safety of AFM11 (Recombinant Antibody Construct Against Human CD19 and CD3) in Patients With Relapsed and/or Refractory CD19 Positive B-cell NHL.
Brief Title: Safety Study to Assess AFM11 in Patients With Relapsed and/or Refractory CD19 Positive B-cell NHL
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Non-favorable risk/benefit profile with studied dosing regimen
Sponsor: Affimed GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AFM11-101; 2013-001919-78 (EudraCT Number)
Record Dates: First submitted 2014-04-01; First posted 2014-04-08 (Estimated); Last update posted 2019-06-18 (Actual); Status verified 2019-05

CONDITIONS: Relapsed B-Cell Non-Hodgkin Lymphoma; Refractory B-Cell Non-Hodgkin Lymphoma
MeSH Terms: conditions — Lymphoma, B-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- AFM11 (Experimental): IV (intravenous) infusion, dose escalation
  Interventions: Drug: AFM11

INTERVENTIONS:
Drug: AFM11 — Accelerated-titration dose-escalation with 1 patient per dose-level, followed by standard dose-escalation (3 + 3 design), Treatment duration: 4 weeks.

SUMMARY:
The purpose of this study is to determine whether AFM11 is safe and active in the treatment of relapsed and/or refractory Non-Hodgkin Lymphoma (NHL).

DETAILED DESCRIPTION:
CD19 is present on B-cells from earliest recognizable B-lineage cells during development to B-cell blasts and is lost only upon maturation to plasma cells. Expression of CD19 on B-cells at various development stages makes it an ideal target to treat B-cell associated malignancies.The rationale for the use of AFM11 is based on its ability to bind to both malignant cells via its anti-CD19 domain and to T-cells via its anti-CD3 domains. This results in the formation of the "immunological synapse" and the subsequent T-cell activation on leading to killing of malignant cells.

ELIGIBILITY:
Inclusion Criteria:

* Patients with CD19+, relapsed or refractory histologically (WHO classification) confirmed follicular lymphoma, marginal zone lymphoma, lymphoplasmocytic lymphoma, mantle cell lymphoma, diffuse large B-cell lymphoma, mediastinal B-cell lymphoma, or transformed B-cell lymphomas.
* Patients with either indolent or aggressive NHL.
* Patients who relapsed or were refractory to the approved standard therapy, which must have included 1 treatment line with rituximab plus chemotherapy, and who are not candidates for bone marrow transplant (including both peripheral blood and hematopoietic stem cell transplants with a curative intent.
* Measurable disease (at least 1 lesion ≥ 1.5 cm) documented by CT scan.
* Disease progression requiring therapy.
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2.
* Life expectancy of at least 6 months.
* Ability to understand the patient information and informed consent form.
* Signed and written informed consent

Exclusion Criteria:

* Total number of B-cells (healthy and malignant combined) in the peripheral blood exceeds the upper physiological limit (as per institutional guidance) of total B-cell counts in healthy individuals.
* Autologous Hematopoietic stem cell transplant (HSCT) within 12 weeks prior to start of AFM11 treatment.
* Abnormal hematological laboratory values as defined below:

  1. Peripheral lymphocyte count > 20 × 10^9/L
  2. Platelet count ≤ 75,000/µL
  3. Hemoglobin level ≤ 9 g/dL.
* Known or suspected central nervous system (CNS) involvement.

  1. History of or current relevant CNS pathology as epilepsy, seizure, paresis, aphasia, apoplexia, severe brain injuries, cerebellar disease, organic brain syndrome, and/or psychosis.
  2. Evidence for presence of malignant disease, inflammatory lesions, and/or vasculitis on cerebral MRI.
  3. Infiltration of the cerebrospinal fluid by malignant B-cells, confirmed by lumbar puncture.
* Cancer chemotherapy within 4 weeks prior to start of AFM11 treatment, or at least 4 times the respective half-lives, whichever is longer.
* Radiotherapy within 4 weeks prior to start of AFM11 treatment.
* Therapy with antibody, or antibody constructs within 4 weeks prior to start of AFM11 treatment, or at least 4 times the respective half-lives, whichever is longer.
* Prior treatment with alemtuzumab (Campath®) within 12 weeks prior to start of AFM11 treatment.
* Treatment with any investigational agent within 4 weeks prior to start of AFM11 treatment, or at least 4 times the respective half-life, whichever is longer.
* Contraindication for any of the concomitant medications.
* Abnormal renal or hepatic function as follows: aspartate aminotransferase (AST or serum glutamic oxaloacetic transaminase [SGOT]) and/or alanine aminotransferase (ALT or serum glutamic pyruvic transaminase [SGPT]) ≥ 2.5 × upper limit of normal (ULN); total bilirubin ≥ 1.5 × ULN; serum creatinine ≥ 2 × ULN; creatinine clearance < 50 mL/minute.
* History of malignancy other than B-cell lymphoma within 5 years prior to study entry, with the exception of basal cell carcinoma of the skin or carcinoma in situ of the cervix.
* Active autoimmune disease requiring systemic immunosuppressive treatment.
* Uncontrolled infections; known bacteremia.
* Any concurrent disease or medical condition that is deemed to interfere with the conduct of the study as judged by the Investigator.
* Regular dose of corticosteroids during the 4 weeks prior to start of AFM11 treatment or anticipated need of continuous corticosteroids exceeding prednisone 20 mg/day or equivalent, or any other immunosuppressive therapy within 4 weeks prior to start of AFM11 treatment.
* Known infection with human immunodeficiency virus (HIV) or chronic infection with hepatitis B or hepatitis C virus.
* Pregnant or nursing women or women of childbearing potential not willing to use an effective form of contraception during participation in the study and at least 12 weeks thereafter. Male patients not willing to ensure that during the study and at least 12 weeks thereafter no fathering takes place. Effective methods of contraception include intrauterine device 8(IUD), combined (estrogen- and progesterone-containing) hormonal contraception (oral, vaginal ring or transdermal patch) with an ethinylestradiol dose of at least 30 µg, plus use of male condoms (preferably with spermicides), female condoms, female diaphragm, or cervical cap.
* Prior treatment with blinatumomab or any other CD19 targeting T-cell engager, including CD19 CAR-T cells.
* Clinically relevant coronary artery disease (New York Heart Association [NYHA] functional angina classification III/IV), congestive heart failure (NYHA III/IV), or high risk of, or known, uncontrolled arrhythmia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2014-04; Primary Completion 2018-08 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Number of participants with serious and non-serious adverse events as a measure of safety and tolerability of AFM11. | From administration of the first dose of study drug and through 30 days after the last dose, up to 8 weeks.
  Measure occurence of adverse events until the Final Study Visit and monitor laboratory safety parameters at least once weekly. Assess immunogenicity of AFM11 at end of treatment cycle.

SECONDARY OUTCOMES:
Maximum Tolerated Dose (MTD) of AFM11. | up to 8 weeks
Pharmacokinetic profile of AFM11 and immunological markers of AFM11 activity. | Prior to initial dose on Day 1 and at multiple time points during the 4 weeks of treatment until up to 30 days after the last dose.
  Concentration of AFM11 in blood samples will measured at different time points during the 4 weeks of treatment and 30 days thereafter to determine concentration-time profiles. Immunological markers like lymphocytes and cytokine levels in serum will be measured at different time points during the 4 weeks of treatment and 30 days thereafter to assess the level of activity resulting from administration of AFM11.
Tumor Response. | Baseline and at week 6.
  Measure tumor size and activity in FDG-PET and CT-scans.

CONTACTS AND LOCATIONS:
Locations (9):
- Tufts Medical Center, Boston, Massachusetts, United States
- Charles Hospital Prague, Prague, Czechia
- Germany (5):
  - University Hospital of the Saarland, Homburg/Saar
  - University Hospital, Kiel
  - University Medical Center of the Johannes Gutenberg University Mainz, Mainz
  - University Hospital, Ulm
  - University Hospital, Würzburg
- Poland (2):
  - SP ZOZ University Hospital Krakow, Krakow
  - MTZ Clinical Research, Warsaw

REFERENCES:
- [Derived] Topp M, Dlugosz-Danecka M, Skotnicki AB, Salogub G, Viardot A, Klein AK, Hess G, Michel CS, Grosicki S, Gural A, Schwarz SE, Pietzko K, Gartner U, Strassz A, Alland L, Mayer J. Safety of AFM11 in the treatment of patients with B-cell malignancies: findings from two phase 1 studies. Trials. 2023 Jan 3;24(1):4. doi: 10.1186/s13063-022-06982-7. PMID 36597128